CLINICAL TRIAL: NCT06819696
Title: A Prospective, Randomized Controlled Study Comparing Tourniquet Use Versus a Dual-flow Arthroscopy Sheath in Anterior Cruciate Ligament (ACL) Reconstruction Surgery.
Brief Title: Tourniquet vs. Dual-flow Arthroscopy Sheath in Anterior Cruciate Ligament (ACL) Reconstruction
Acronym: RELICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-CHITS-007; 2024-A01117-40 (Other: ID-RCB number)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior Cruciate Ligament; Arthroscopy; Dual-flow arthroscopy sheath; Tourniquet; pain; Surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will be masked to the surgical procedure and will be unblinded upon completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-flow arthroscopy sheath (Experimental): Patients will undergo ACL reconstruction using a dual-flow arthroscopy sheath.
  Interventions: Procedure: ACL reconstruction with a dual-flow arthroscopy sheath
- Thigh tourniquet (Active Comparator): Patients will undergo ACL reconstruction using a thigh tourniquet.
  Interventions: Procedure: ACL reconstruction with a thigh tourniquet

INTERVENTIONS:
Procedure: ACL reconstruction with a dual-flow arthroscopy sheath — ACL reconstruction will be performed by the surgeon without a tourniquet but using a dual-flow arthroscopy sheath.
  Arms: Dual-flow arthroscopy sheath
Procedure: ACL reconstruction with a thigh tourniquet — ACL reconstruction will be performed by the surgeon using a thight tourniquet
  Arms: Thigh tourniquet

SUMMARY:
This is a prospective randomized study comparing tourniquet use versus a dual-flow arthroscopy sheath in Anterior Cruciate Ligament (ACL) reconstruction surgery.

The ACL is largely responsible for knee stability and contributes to central pivot with the posterior cruciate ligament. ACL rupture is associated with a violent twisting motion of the knee, which is usually irreparable without surgical intervention.

ACL reconstruction via arthroscopy is the gold standard treatment for young, active patients with knee instability. Reconstruction is commonly performed using a thigh tourniquet to improve intraoperative visibility, reduce bleeding, and shorten procedure time. However, numerous studies associate tourniquet use with an increased risk of postoperative complications such as increased pain, muscle injury, postoperative bleeding, and deep vein thrombosis. Therefore, it seems relevant to conduct further investigations into the benefits of new methods to replace tourniquet. In this context, the dual-flow arthroscopy sheath could improve postoperative recovery after ACL reconstruction and could limit the risk of complications, thus improving ambulatory care for patients.

This study propose to compare two groups of patients undergoing ACL reconstruction: those operated on with a tourniquet versus those operated on using the dual-flow arthroscopy sheath.

DETAILED DESCRIPTION:
Initial assessments will be conducted preoperatively. The follow-up examination will take place during the first 7 days following surgery and then at 21 days (D21), 45 days (D45), and 5 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Primary ACL reconstruction
* Age 18 years or older
* Provided informed consent prior to study participation
* Affiliated to or beneficiary of a social security regimen

Exclusion Criteria:

* Multi-ligamentous surgery
* Revision ACL surgery
* Presence of a meniscal and/or chondral lesion not allowing immediate weight-bearing postoperatively
* Bleeding disorder
* Pregnant, parturient or breastfeeding women
* Patient under legal guardianship
* Any other reason which, in the opinion of the investigator, could interfere with the evaluation of the objectives of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity according to a Numeric Rating Scale (NRS) | 4 days after surgery
  Pain intensity will be assessed using a Numeric Rating Scale (NRS) at 8 AM, 12 PM, and 8 PM on postoperative day 4.
  The minimum value of the scale, corresponding to no pain at all, is 0 and the maximum value is 10.

SECONDARY OUTCOMES:
Pain intensity according to a Numeric Rating Scale (NRS) | Up to 3 days after surgery
  Pain intensity will be assessed using a Numeric Rating Scale (NRS) on the day of surgery (preoperatively and at 4, 12, and 16 hours postoperatively) and on days 1, 2, and 3 following surgery (at 8 AM, 12 PM, and 8 PM).
  The minimum value of the scale, corresponding to no pain at all, is 0 and the maximum value is 10.
Total antalgic consumption | Up to 4 days after surgery
  Total antalgic consumption will be assessed in number of doses per type of drug, from surgery up to 4 days after surgery.
Arthrogenic Muscle Inhibition (AMI) classification | Preoperative, on Day 0 before and after surgery and then on Day 21 and Day 45 after surgery.
  This classification is used to assess quadriceps contraction.
Lysholm knee scoring scale | Preoperative, Day 21, Day 45 and Month 5 after surgery
  The Lysholm Knee Score is a standardized questionnaire used to assess knee function after surgery. The total score obtained ranges from 0 to 100. The higher the score, the better the knee's function.
Knee Blessure and Osteoarthritis Outcomescore (KOOS) | Preoperative, Day 21, Day 45 and Month 5 after surgery
  The KOOS is a self-administered questionnaire that evaluates multiple aspects of knee health, including pain, symptoms, daily living activities, sports and recreation function, and quality of life.
  Each subscale is rated from 0 to 100, where 0 represents extreme problems and 100 represents no problem.
Knee mobility | Preoperative, Day 21, Day 45 and Month 5 after surgery
  Knee mobility will be assessed using a goniometer.
Total surgical time | Day 0
  Assessed in minutes
Arthroscopic time | During procedure
  Assessed in minutes
Intraoperative visibility | During procedure
  Intraoperative visibility will be assessed by the surgeon using a 4-point scale (excellent, good, fair, poor).
Thigh, knee and calf diameters in cm | Preoperative and Day 21
  Diameters will be evaluated in cm.
CPK blood level | Preoperative and Day 1
Hemoglobin level | Preoperative, Day 1 and Day 7
Presence of complications | Up to 5 months
  The number and type of complications will be recorded, including hematomas, knee stiffness, deep vein thrombosis, complex regional pain syndrome, deep infection, superficial infection, and recurrent anterior cruciate ligament graft rupture.
Muscle strength | Preoperative and 5 months
  Muscle strength will be assessed in both limbs using isokinetic testing

CONTACTS AND LOCATIONS:
Overall Officials: Cédric SIEDLECKI, MD, Study Director — Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer and Centre Hospitalier de Hyères
Locations (2):
- France (2):
  - Centre Hospitalier de Hyères, Hyères, Var
  - Centre Hospitalier Intercommunal Toulon - La Seyne sur Mer, Toulon, Var

IPD SHARING:
Plan to Share IPD: No